CLINICAL TRIAL: NCT05911802
Title: Prognostic Analyses on a Validation Series of Patients With Waldenström's Disease: Validation of International Prognostic Indexes, Evaluation of Progression-free Survival as a Surrogate Endpoint for Overall Survival. A FILO Study.
Brief Title: Prognostic Analyses on a Validation Series of Patients With Waldenström's Disease
Acronym: SérieProWM
Status: Recruiting | Type: Observational
Sponsor: French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Other Study IDs: FILObs_SérieProWM
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Waldenstrom's Disease; Prognostic Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — bone marrow samples for analysis like genetic analysis (MYD88 (L265P) and CXCR4 mutational status)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- symptomatic WM: WM patients with symptom(s) : cytopenia, bulky disease or when the physicochemical or immunological properties of IgM explain the occurrence of amyloidosis, cryoglobulin, neurological manifestations, or hyperviscosity syndrome (due to the presence of a large amount of IgM)
- asymptomatic WM: WM patients without any symptom

SUMMARY:
Waldenström's macroglobulinemia (WM) is defined by the association of bone marrow lymphoplasmocytic infiltration and monoclonal immunoglobulin M (IgM). A mutation in the MYD88 gene is found in up to 90% of patients, and a mutation in the CXCR4 gene in approximately one third of patients. Treatment should be initiated in cases of cytopenia, bulky disease or when the physicochemical or immunological properties of IgM explain the occurrence of amyloidosis, cryoglobulin, neurological manifestations, or hyperviscosity syndrome (due to the presence of a large amount of IgM). However, approximately 30% of patients are diagnosed without any symptom and therefore they do not meet the criteria for initiating treatment.

At the time of initiation of the first treatment, the prognosis is usually estimated with the International Prognostic Index (IPSSWM) which is based on five variables: age, platelet count, haemoglobin concentrations, β2-microglobulin and monoclonal component concentration. Serum albumin and lactate dehydrogénase (LDH) levels also retain a prognostic role and these two characteristics have been incorporated in a proposal for a revision of this index.

Improving prognostic assessment at the time of the first treatment initiation and taking into account the prognostic impact of events occurring in the course of evolution, should improve the strength of treatment decision at the time of initial treatment and during the follow-up. It should also help to design clinical trial for fast and effective evaluation of new treatments. Our work should also help to adjust clinical monitoring of asymptomatic patients.

Prospective and retrospective multicenter prognostic study with a descriptive objective, associated with a biological collection appropriately annotated and stored. A retrospective series including 470 patients with symptomatic WM is already available. The follow-up of these patients will be updated and an additional series of 250 symptomatic patients will be prospectively enrolled. 250 asymptomatic patients will be also enrolled.

DETAILED DESCRIPTION:
Waldenström's macroglobulinemia (WM) is defined by the association of bone marrow lymphoplasmocytic infiltration and monoclonal immunoglobulin M (IgM). A mutation in the MYD88 gene is found in up to 90% of patients, and a mutation in the CXCR4 gene in approximately one third of patients. Treatment should be initiated in cases of cytopenia, bulky disease or when the physicochemical or immunological properties of IgM explain the occurrence of amyloidosis, cryoglobulin, neurological manifestations, or hyperviscosity syndrome (due to the presence of a large amount of IgM). However, approximately 30% of patients are diagnosed without any symptom and therefore they do not meet the criteria for initiating treatment.

The prognosis of asymptomatic patients can be estimated with a prognostic index based on serum albumin, β2-microglobulin, the monoclonal component concentration and the bone marrow infiltration. Prognostic assessment of these patients could be improved by taking into account prior the free light chain concentrations and the molecular characteristics of the disease.

At the time of initiation of the first treatment, the prognosis is usually estimated with the International Prognostic Index (IPSSWM) which is based on five variables: age, platelet count, haemoglobin concentrations, β2-microglobulin and monoclonal component concentration. Serum albumin and LDH levels also retain a prognostic role and these two characteristics have been incorporated in a proposal for a revision of this index.

Thus improving prognostic assessment in patients with WM may rest on the following strategies:

* Modifying the variables to be considered before treatment initiation, particularly by considering albumin and lactate dehydrogenase concentrations or molecular characteristics of the disease in symptomatic patients, free-light chain concentration in asymptomatic patients and molecular abnormalities in both categories of patients.
* Evaluating the prognostic impact of events occurring during the course of treatment, such as response or progression in symptomatic patients.

Improving prognostic assessment at the time of the first treatment initiation and taking into account the prognostic impact of events occurring in the course of evolution, should improve the strength of treatment decision at the time of initial treatment and during the follow-up. It should also help to design clinical trial for fast and effective evaluation of new treatments. Our work should also help to adjust clinical monitoring of asymptomatic patients.

Two large subgroups of patients properly included with validated information and updated follow-up will be considered, namely: symptomatic and asymptomatic patients. This project is based on the assumption that it should be possible for each of these two cohorts to:

1. validate a new prognostic system and compare its performance with previous systems
2. to participate in a large international study of the validity of a surrogate endpoint of survival after initiation of the 1st treatment

ELIGIBILITY:
Inclusion Criteria:

* Patient with WM, fulfilling the diagnostic criteria defined at the 2nd Workshop on WM.
* Patient in whom follow-up is available until at least 01/01/2020. Each participating center should not enroll more 10% of patients lost to follow-up.
* Patient for whom a minimum annual follow-up is planned until 2024.
* Having given their consent for this study

Exclusion Criteria:

* Patient with other chronic lymphoid malignancy. Special attention will be paid to exclude other lymphoplasmacytic proliferations, especially marginal zone lymphoma.
* Patient with histological transformation in a diffuse large B-cell lymphoma or any other lymphoma at the time of the initiation of the 1st treatment.
* No consent for this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 250 symptomatic patients and 250 asymptomatic patients will be prospectively enrolled
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2030-06-15 (Estimated); Study Completion 2030-06-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years after WM diagnosis
  Percentage of living patients

SECONDARY OUTCOMES:
Progression free survival | 1 year after WM diagnosis
  percentage of living patients without disease progression
Tolerance to treatment | 1 year after initiating WM treatment
  percentage of patients discontinuing WM treatment due to toxicity

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - AMIENS - CH Amiens Picardie Site Sud, Amiens
  - Angers Chu, Angers
  - Institut Bergonie, Bordeaux
  - Clermont-Ferrand - Chu Estaing, Clermont-Ferrand
  - Le Mans CH, Le Mans
  - LENS - GHT Artois, Lens
  - LIBOURNE - Hôpital Robert Boulin, Libourne
  - LILLE GHICL - Hôpital Saint Vincent de Paul, Lille
  - Institut Paoli Calmette, Marseille
  - APHP - Hôpital Pitié Salpêtrière - Hématologie, Paris
  - POITIERS - Hématologie et Thérapie Cellulaire, Poitiers
  - Reims Chu, Reims
  - Strasbourg - Icans, Strasbourg
  - Toulouse - IUCT Oncopole - Service d'Hématologie, Toulouse
  - VERSAILLES - Hôpital André Mignot, Versailles

IPD SHARING:
Plan to Share IPD: Undecided
Specific or all individual participant data sets would be probably shared with the European ECWM Group. For example, data on use of BTKi ( Bruton tyrosine kinases inhibitors) in this population

REFERENCES:
- [Background] Royston P, Altman DG. External validation of a Cox prognostic model: principles and methods. BMC Med Res Methodol. 2013 Mar 6;13:33. doi: 10.1186/1471-2288-13-33. PMID 23496923